CLINICAL TRIAL: NCT01915901
Title: A Multicenter, Double Blind, Placebo-Controlled Study of Pepto-Bismol® (Bismuth Subsalicylate) on Gastrointestinal Tolerability in Healthy Volunteers Receiving Oral TECFIDERA™ (Dimethyl Fumarate) Delayed-Release Capsules Twice Daily
Brief Title: PeptoBismol® Use to Reduce Gastrointestinal Events in Healthy Volunteers Receiving DMF [Tecfidera®] Twice Daily
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109HV110
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
MeSH Terms: interventions — bismuth subsalicylate; Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- bismuth subsalicylate (Pepto-Bismol®) + DMF (Experimental): Subjects will receive dimethyl fumarate (DMF) and bismuth subsalicylate (Pepto-Bismol®).
  Interventions: Drug: bismuth subsalicylate (Pepto-Bismol®); Drug: dimethyl fumarate (DMF)
- Placebo + DMF (Experimental): Subjects will receive dimethyl fumarate (DMF) and placebo.
  Interventions: Drug: matching placebo (bismuth subsalicylate); Drug: dimethyl fumarate (DMF)

INTERVENTIONS:
Drug: bismuth subsalicylate (Pepto-Bismol®) — 524 mg bismuth subsalicylate twice a day (BID)
  Other Names: Pepto-Bismol®
  Arms: bismuth subsalicylate (Pepto-Bismol®) + DMF
Drug: matching placebo (bismuth subsalicylate) — placebo twice a day (BID)
  Arms: Placebo + DMF
Drug: dimethyl fumarate (DMF) — dimethyl fumarate (DMF) twice a day (BID)
  Other Names: BG00012; DMF; TECFIDERA™

SUMMARY:
The primary objective of the study is to determine the effect of bismuth subsalicylate (Pepto-Bismol®) 524 mg versus placebo on gastrointestinal (GI)-related events reported in healthy volunteers receiving TECFIDERA™ (dimethyl fumarate [DMF]; also known as BG00012) twice daily (BID) The secondary objectives of this study in this study population are: To characterize the effect of bismuth subsalicylate (Pepto-Bismol®) 524 mg versus placebo on the frequency, severity, and duration of GI-related events and to evaluate GI-related events that lead to discontinuation of DMF.

ELIGIBILITY:
Key Inclusion Criteria:

* Must be in good health as determined by the Principal Investigator (PI) based on medical history and Screening evaluations (clinical laboratory evaluations, 12-lead electrocardiogram (ECG), and vital signs; see below for specific exclusion criteria).
* Must have a body mass index (BMI) of 18.0 to 34.0 kg/m2, inclusive.
* Subjects of reproductive potential (including males) must practice effective contraception during the study and be willing and able to continue contraception for 90 days after their last dose of study drug.
* Male subjects must agree to not donate sperm for 90 days after their last dose of study drug.
* Must be naïve to dimethyl fumarate (DMF) or fumaric acid esters.

Key Exclusion Criteria:

* History of or positive results at the Screening visit for HIV.
* History of or positive results at the Screening visit for hepatitis C virus antibody or hepatitis B virus (defined as positive for hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb]).
* History of clinically significant gastrointestinal (GI) disease as determined by the PI (including Crohn's disease, peptic ulcer disease, ulcerative colitis, or confirmed diagnosis of irritable bowel syndrome) or active GI disease with ongoing symptoms.
* History of severe allergic or anaphylactic reactions, considered clinically relevant by the PI.
* Known allergy to Pepto-Bismol®, salicylates, or non-steroidal anti-inflammatory drugs, considered clinically relevant by the PI.
* Female subjects who are pregnant based on results of the serum pregnancy test at Screening or currently breastfeeding.
* Current enrollment in any other study treatment or disease study.
* Receipt of any investigational drug within 5 half-lives or 30 days, whichever is longer, prior to study entry.
* History of alcohol abuse or substance abuse (as determined by the PI) within the previous 5 years, a positive urine drug/alcohol test at Screening, or alcohol use prior to the screening visit.
* Regular use of any tobacco product, defined as smoke or smokeless product use equivalent to >5 cigarettes/day for any consecutive week, within 3 months prior to Day 1.

Other unspecified reasons that, in the opinion of the PI or Biogen Idec, make the subject unsuitable for enrollment.

Other protocol-defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Time to first gastrointestinal-related event | Up to 8 weeks

SECONDARY OUTCOMES:
The number of gastrointestinal-related events. | Up to 8 weeks
The duration of gastrointestinal-related events. | Up to 8 weeks
The severity of gastrointestinal-related events. | Up to 8 weeks
The percentage of subjects who discontinue dimethyl fumarate (DMF) due to gastrointestinal-related events | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (3):
- United States (3):
  - Research Site, Daytona Beach, Florida
  - Research Site, Dallas, Texas
  - Research Site, Madison, Wisconsin

REFERENCES:
- [Derived] Koulinska I, Riester K, Chalkias S, Edwards MR. Effect of Bismuth Subsalicylate on Gastrointestinal Tolerability in Healthy Volunteers Receiving Oral Delayed-release Dimethyl Fumarate: PREVENT, a Randomized, Multicenter, Double-blind, Placebo-controlled Study. Clin Ther. 2018 Dec;40(12):2021-2030.e1. doi: 10.1016/j.clinthera.2018.10.013. Epub 2018 Nov 15. PMID 30447891